CLINICAL TRIAL: NCT01963767
Title: Phase II Study of a Nutraceutical on the Cognitive Performance of Older Adults.
Brief Title: Nutraceutical Effects on Long-Term Memory
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Pro00001021; 24127 (Other Grant/Funding Number: University of South Florida)
Record Dates: First submitted 2013-10-09; First posted 2013-10-16 (Estimated); Results first posted 2014-07-04 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-04

CONDITIONS: Aging
Keywords: memory; cognition; dietary supplements
MeSH Terms: interventions — NT020 formula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NT-020 (Experimental): Participants received two pills of NT-020 plus Biovin (900 mg proprietary formulation of blueberry, carnosine, green tea, plus 200 U Vitamin D3, 40 mg Biovin), with one to be taken in the morning and the other in the evening.
  Interventions: Drug: NT-020
- Placebo (Placebo Comparator): Subjects took two pills, one in the morning and one in the evening, that were matched in size and shape to the active compound.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Drug: NT-020 — Recommended intake of NT-020 (NutraStem®) is two (2) capsules daily. This comprises Vitamin D3 (2000 IU), BioVin® (40 mg) and the proprietary blend (900mg). This recommended intake was calculated from doses analyzed in scientific research and based on the dose within the submitted patent.
  Scientific description of the ingredients of the product per a 2 capsule dose Vitamin D3 (as cholecalciferol) - 2000 IU BioVin® Grape Extract - 40 mg Proprietary Blend - 900mg Green Tea Extract (Camellia sinensis) Wild Blueberries* (whole fruit) Carnosine VitaBlue® Wild Blueberry Extract*
  * Vaccinium angustifolium
  Other Ingredients:
  Magnesium stearate, Cellulose (vegetarian capsules) Contains no yeast, wheat, corn, milk, egg, soy, glutens, artificial colors or flavors, added sugar, starch or preservatives.
  Other Names: Naturatherapeutics Nutrastem
  Arms: NT-020
Dietary Supplement: Placebo
  Other Names: Participants were to take two placebo pills, one in the morning and one at dinner.
  Arms: Placebo

SUMMARY:
Interventions to improve the cognitive health of older adults are of critical importance. In the current protocol, ithe investigators conducted a short-term (two months) randomized clinical trial to examine the influence of the nutraceutical NT-020 on the cognitive performance of older adults. Participants were tested with a battery of cognitive tasks at baseline and two months after being randomized to the interventional drug or placebo.

DETAILED DESCRIPTION:
SUMMARY OF STUDY PLAN

The proposed clinical study is a Phase II, randomized, double-blinded, placebo-controlled trial in adults 65-85 years of age with no evidence of cognitive impairment. A total of 120 persons will be randomized to the study, with the goal of completing 100 evaluable subjects.

At the screening assessment, participants will complete the informed consent; questionnaires on basic demographic information including personal medical history and allergies to drug compounds; a mental ability test called the Mini-Mental Status Examination (MMSE); the SF-12 Health survey; the Centers for Epidemiologic Studies Depression Scale (CES-D) and distribute instructions and forms for diet survey and gastrointestinal questionnaires.

At the baseline/randomization assessment, study staff will (a) Confirm eligibility based on screening tests; (b) collect completed diet and gastrointestinal questionnaire survey forms; (c) collect blood for CBC/CMP and antioxidant biomarkers; (d) battery of cognitive tests including Rey Auditory Verbal Learning Test, Educational Testing Service - Identical Pictures Test, Educational Testing Service - Number Comparison Test, Educational Testing Service - Vocabulary Test, Trailmaking A & B, Wechsler Adult Intelligence Scale - Digit Symbol Test, Wechsler Intelligence Scale - Digit Span, Letter Fluency, Category Fluency. Subjects will be equally randomized (n=60 per arm) to blinded treatment with either NT-020 (Natura Therapeutics Nutrastem) or matching placebo, and an initial supply of study drug will be dispensed. Participants will be supplied with one-month supply of blinded treatment (n=60/arm) and be given the study agent intake and symptom log form. The planned intervention period is 2 months.

At specified intervals (weeks 1, 3, 5, 7), participants will be contacted to inquire about the correct administration of the supplement or placebo as well as to assess for any adverse events.

At one month (midpoint), participants will return to campus to (a) collect blood for CBC/CMP and antioxidant biomarkers, (b) collect unused nutritional supplement or placebo and completed study agent intake and symptom log form; (c) collect completed diet survey; (d) supply participant with new one-month supply of nutritional supplement or placebo and new study agent intake and symptom log form.

At the end of the intervention (2 months), we will (a) collect blood for CBC/CMP and antioxidant biomarkers; (b) collect unused nutritional supplement or placebo and completed study agent intake and symptom log form; (c) collect completed diet survey; (d) battery of cognitive tests including Rey Auditory Verbal Learning Test, Educational Testing Service - Identical Pictures Test, Educational Testing Service - Number Comparison Test, Educational Testing Service - Vocabulary Test, Trailmaking A & B, Wechsler Adult Intelligence Scale - Digit Symbol Test, Wechsler Intelligence Scale - Digit Span, Letter Fluency, Category Fluency; ; (e) complete eyeblink conditioning paradigm; (f) complete timed interval tapping paradigm; and (g) Memory Abilities Questionnaire (MAQ-SR);

The primary endpoint of the study is a comparison of the delay eyeblink acquisition performance between persons in the placebo and intervention arms. Other endpoints include: assessing the safety of NT-020 under the proposed dosing regimen; investigating the effect of NT-020 on additional measures of cognitive performance. An additional exploratory endpoints is to examine results from serum and urine diagnostic markers (C-reactive protein, IL-1B, TNFa) after 2 months of intervention with nutritional supplement vs. placebo.

STATISTICAL CONSIDERATIONS

Study Design/Endpoints

The central hypothesis for this Phase II clinical trial is that adults who receive NT-020 will exhibited faster acquisition of the delay eyeblink conditioning, as compared to adults on the placebo.

Sample Size/Accrual Rate We anticipate screening 120 persons, randomizing 100, and having 88 persons complete the two-month study period. We powered the analysis for the repeated measures ANOVA for the eyeblink conditioning paradigm. Power was estimated to be .80 (α = .05), assuming six blocks of trials during the acquisition of the CR, an effect size of f = .16 for the group X trials interaction, and a sample size of 44 per group, assuming an attrition rate of 12% over the two month period.

Randomization and Stratification During the baseline/randomization visit, subjects will be randomized using the stratified randomization method prior to intervention by utilizing a web-based randomization system.

Primary Endpoints The primary efficacy endpoint is to compare the acquisition of delay eyeblink conditioning between persons treated with NT-020 vs. placebo. The planned intervention period is two months. Eyeblink conditioning outcomes will be examined using a 2 (group; NT-020, placebo) X 6 (trial) repeated measures ANOVA to examine differences in the acquisition of the conditioned response from the eyeblink conditioning.

Secondary Endpoint(s) Is the facilitation of the acquisition of the delay and trace human eyeblink response in the nutritional supplementation group mediated by changes in anti-oxidant markers? In order to examine the mediation of the intervention group effects on eyeblink acquisition, we will adopt Baron and Kenny's approach to regression-based statistical mediation. In this model, there are several requirements that must be satisfied in order to claim statistical mediation. We will examine whether intervention group is associated with eyeblink acquisition, whether intervention group is associated with changes in biomarkers, as well as the critical step of whether the influence of intervention group on eyeblink acquisition is reduced or made not statistically significant by the inclusion of changes to biomarker values in the regression analysis.

Evaluate the effect of NT-020 treatment on changes in paper and pencil measures of cognitive performance: A 2 (time; baseline, two-months) X 2 (group; NT-020, placebo) ANOVA will be computed on each of the cognitive test scores. The presence of a group X time interaction will suggest that the two groups exhibit differential change across the two time points.

ELIGIBILITY:
Inclusion Criteria:

* Adults 65-85 years of age (inclusive).
* Able to understand and sign the informed consent.
* Native English-speaking.
* No evidence of dementia (MMSE >=23).
* Each subject must be willing to give consent after being informed of the experimental nature of therapy, alternatives, potential benefits, side-effects, risks and discomforts.
* All subjects must be willing to be monitored for adequacy of nutritional intake during the intervention, as is the current standard of clinical practice.

Exclusion Criteria:

* Use of high dose antioxidant supplements other than what is provided in the trial.
* History of known allergy to components of the study supplements.
* Mental illness judged by the PI to preclude a successful completion of the trial.
* Persons who are not native English speakers are excluded from the current proposal because many of the cognitive tests that are administered are language-based and are heavily influenced by first language.
* Other acute or chronic medical or psychiatric condition or laboratory abnormality that may increase risk associated with study participation or study drug administration, or may interfere with interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 139 (Actual)
Dates: Start 2011-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brent J Small, PhD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: From the 139 participants who were consented in the study, only 113 participated in the baseline assessment. Of the 26 who did not participate in the baseline assessment, 14 failed the screening and 12 dropped out before the baseline assessment.
Groups:
- NT-020: Participants received two pills of NT-020 plus Biovin (900 mg proprietary formulation of blueberry, carnosine, green tea, plus 200 U Vitamin D3, 40 mg Biovin), with one to be taken in the morning and the other in the evening.
  NT-020: Recommended intake of NT-020 (NutraStem®) is two (2) capsules daily. This comprises Vitamin D3 (2000 IU), BioVin® (40 mg) and the proprietary blend (900mg). This recommended intake was calculated from doses analyzed in scientific research and based on the dose within the submitted patent.
Period: Overall Study
Arm/Group | NT-020 | Placebo
Started | 58 | 55
Completed | 52 | 53
Not Completed | 6 | 2
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Population: Description is limited to persons who completed the entire study. The eight subjects who did not complete the study are excluded from this table.
Groups:
- Total: Total of all reporting groups
Arm/Group | NT-020 | Placebo | Total
Number analyzed (Participants) | 53 | 52 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.34 (5.48) | 72.82 (5.54) | 73.58 (5.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 33 | 65
  Male | 21 | 19 | 40
Years of Education [Mean (Standard Deviation); unit: years] | 15.61 (2.93) | 15.88 (2.41) | 15.75 (2.67)

OUTCOME MEASURES:

1. Primary Outcome: Delay Eyeblink Conditioning
Description: Participants will be tested on eyeblink classical conditioning at the USF Health Byrd Alzheimer's Institute. Participants will receive 60 trials of eyeblink conditioning at the two-month follow-up point. Participants watch an entertaining silent video (e.g., Milo and Otis). The airpuff is delivered through a nozzle held in front of the participant and blink latency is recorded.
  The outcome measure is an index of the percentage of eyeblinks that are made to a tone (conditioned stimulus) after the learning period is complete. The percentage can range from 0% (no conditioned learning has occurred) to 100% (all responses are conditioned; Woodruff-Pak, D. S. (2001). Eyeblink classical conditioning differentiates normal aging from Alzheimer's disease. Integrative Physiological and Behavioral Science, 36(2), 87-108.).
Time Frame: Measured at the end of the intervention period, which is two months after initiation of the placebo of NT-020 doses
Population: From the 105 persons with complete data on the second outcome, only 102 had complete data on this outcome. The three who did not contribute to this analysis were because there were two equipment failures and one person had a glass eye and the procedure could not be performed.
Measure: Mean (Standard Deviation); unit: percentage of conditioned responses
Groups:
- NT-020: Participants received two pills of NT-020 plus Biovin (900 mg proprietary formulation of blueberry, carnosine, green tea, plus 200 U Vitamin D3, 40 mg Biovin), with one to be taken in the morning and the other in the evening.
  NT-020: Recommended intake of NT-020 (NutraStem®) is two (2) capsules daily. This comprises Vitamin D3 (2000 IU), BioVin® (40 mg) and the proprietary blend (900mg). This recommended intake was calculated from doses analyzed in scientific research and based on the dose within the submitted patent.
  Scientific description of the ingredients of the product per a 2 capsule dose Vitamin D3 (as cholecalciferol) - 2000 IU BioVin® Grape Extract - 40 mg Proprietary Blend - 900mg Green Tea Extract (Camellia sinensis) Wild Blueberries* (whole fruit) Carnosine VitaBlue® Wild Blueberry Extract*
  * Vaccinium angustifolium
Arm/Group | NT-020 | Placebo
Number analyzed (Participants) | 50 | 52
percentage of conditioned responses | 52.32 (26.85) | 56.88 (28.42)

2. Secondary Outcome: Cognitive Performance
Description: The secondary endpoint will be improvement in cognitive performance over the two-month follow-up period on the paper and pencil tests of cognitive ability. The test that was used here is the Identical Pictures test, from the Educational Testing Services battery (Ekstrom RB, French JW, Harman HH, Dermen D. Manual for kit of factor referenced cognitive tests. Educational Testing Service, Princeton, NJ, 1976.). This test evaluates the number of pictures that persons can match within a 90 second period. There are two trials at 90 seconds and the maximum score is 48 matches (minimum is 0). Higher scores indicate better performance because participants are able to make more matches within the 90 second interval. This test provides an index of processing speed, the ability to do a task rapidly.
Time Frame: Measured at baseline and two months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | NT-020 | Placebo
Number analyzed (Participants) | 52 | 53
units on a scale | 24.12 (.65) | 21.72 (.61)
Statistical Analysis 1: Comparison: NT-020 vs Placebo; Ancovas were conducted with group as the between subjects factor and performance at baseline as the covariate; Test type: Superiority or Other; p = .03, ANCOVA

ADVERSE EVENTS:
Arm/Group | NT-020 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/52 | 0/53
Other Adverse Events (participants affected / at risk) | 2/52 | 1/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NT-020 (N=52) | Placebo (N=53)
Cardiac disorders (Cardiac disorders) | 1 (1) | 0 (0) — One participant exhibited a significant cardiac adverse event during the course of the study during her first month of participation. This event was reported to Western IRB and it was determined to be unrelated to her participation in the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NT-020 (N=52) | Placebo (N=53)
Upset Stomach (Gastrointestinal disorders) | 2 (2) | 1 (1) — Some participants complained of an upset stomach while taking the compounds

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No